CLINICAL TRIAL: NCT03038685
Title: A Personalized, Digital Coaching Program With Teleconsultancy to Improve Secondary Prevention After Ischemic Stroke: a Pilot, Multicenter Pre/Post Study.
Brief Title: A Personalized, Digital Coaching Program After Stroke
Acronym: STROKECOACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Sint-Lucashospital, Bruges, Belgium (Unknown); AZ Sint-Jan AV (Other); Groeningehospital, Kortrijk, Belgium (Unknown); Belgian Stroke Council (Unknown); Interuniversity Centre For Health Economics Research, VUB, Brussels, Belgium (Unknown)
Responsible Party: Principal Investigator, PVanacker, neurovascular consultant, University Hospital, Antwerp
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UHAntwerp
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Stroke, Ischemic
Keywords: Secondary prevention; Web-based intervention; Strokecoach
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: A pilot, double-arm, pre/post study design with compirason between historical, monocenter cohort (Sint-Janhospital, 2011) and prospective, multicenter cohort (4 Belgian Stroke centers, 2017)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prospective, multicenter cohort (Experimental): A group of 175 patients will be recruited in 4 Belgian stroke centers during the six months period. All data will be collected prospectively and patients will be treated during six months period.
  Interventions: Behavioral: Strokecoach.be - digital coaching program for stroke patients
- historical, single center cohort (No Intervention): A historical cohort of Sint-Janhospital (2011 - Bruges, Belgium) with prospectively collected data will be used as comparator for the experimental arm. These data were published in Vanacker P, Couvreur T, Vanhooren G. Can we improve cerebrovascular risk reduction in real-life? A single centre's experience. Cerebrovasc Dis 2011;31(suppl 2):289

INTERVENTIONS:
Behavioral: Strokecoach.be - digital coaching program for stroke patients — The stroke coach gives patients two education sessions during hospitalization (risk factor management, review of medications and clinical evolution). During these sessions, study participation will be proposed. Eligibility will partially depend on their historical use of the internet and e-mail. The aim is to have the digital platform personalized for his/her individual needs, risk factors and remaining neurologic signs/symptoms. Tips and tricks to deal with lifestyle modification will be delivered on regular basis. Meanwhile, patients will be asked to complete on a pre-specified frequency their data regarding their cardiovascular risk profile. Additionally, participants will be contacted at 0.5-1-2 and 6 months by phone calls or videoconsultancy. To standardize, an adapted, digital version of the standardized WSO Post-Stroke Checklist shall be used as a decision-support flowchart. A report of the consultation will be derived after the videoconsultancy.
  Arms: prospective, multicenter cohort

SUMMARY:
The Belgian Stroke Council initiated a project to improve risk factor control and medication adherence in ischemic stroke patients by developing an individualized in-hospital initiated and post- discharge, digital coaching program addition to standard practice (strokecoach.be).

DETAILED DESCRIPTION:
The overall aim of this project is to further improve subacute and chronic stroke care in the Belgian context with main focus on the patients' quality of life, stroke recurrence and secondary cardiovascular prevention. Main focuses are on patient-empowerment, shared-decision making and health literacy, as these items are linked with better therapeutic adherence and self-care for chronic diseases.

In case of a positive result, implementation of this individualized chronic stroke care program executed by a personal stroke coach, initiated during hospitalization and using a web-based intervention program, can easily be unrolled in other Belgian stroke units. The program can be cost-effective if better clinical outcome, stroke recurrence rates, number of in-hospital consultations, number of rehospitalisations are reduced. This will be evaluated in a in-depth healt-economic analysis.

ELIGIBILITY:
Inclusion Criteria:

Patients with an acute ischemic stroke hospitalized at a participating stroke center can be included during hospitalisation if fulfilling following three criteria: - they will return back home or be discharged to a rehabilitation center

* have a life expectancy of more than 6 months
* have experience with internet use (at least weekly checking emails) or a caregiver accepts to help with the digital platform.

Exclusion Criteria:

* Age < 18 years
* Patients unable or unwilling to be followed post-discharge for 6 months
* Patients with a major neurologic post-stroke and no caregiver participation
* Cognitive impairment limiting use of digital platform and no caregiver participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
cardiovascular risk factor control | 6 months
  The primary endpoint is the impact of the intervention on the cardiovascular risk factor control by assessing the evolution of the SCORE (Systematic COronary Risk Evaluation: High & Low cardiovascular Risk Charts) risk pre- and postintervention. An official program to analyze these parameter will be used (AOST©, Crethsoft).

SECONDARY OUTCOMES:
Quality-of-life | 3-6months
  The impact on the quality-of-life will be evaluated by using the dutch version of the EQ-5D questionnaire
Clinical outcome | 6 months
  The impact on the clinical outcome will be assessed by the modified Rankin Score (0-6, mRS).
Stroke recurrence rate | 0.5-1-2-3-6 months
  At every teleconsultancy contact stroke recurrences will be demanded.
Therapeutic adherence | 0.5-1-2-3-6 months
  A selfreport of the therapeutic adherence will be checked at every consultation by asking them if any medication had been skipped during last 10 days.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vanacker, MD PhD, Principal Investigator — University Hospital, Antwerp
Locations (4):
- Belgium (4):
  - Sint-Janhospital, Bruges
  - Sint-Lucashospital, Bruges
  - University Hospital Antwerp, Edegem
  - Groeningehospital, Kortrijk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31701472/